CLINICAL TRIAL: NCT06191094
Title: A Randomized, Double-masked, Sham-controlled Study to Evaluate the Efficacy of Peri-operative Farcimab in Patients With Non-clearing Vitreous Hemorrhage Secondary to Proliferative Diabetic Retinopathy
Brief Title: Pre-operative Vabysmo in Patients With Non-clearing Vitreous Hemorrhage Secondary to Proliferative Diabetic Retinopathy
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 23-0483
Record Dates: First submitted 2023-12-08; First posted 2024-01-05 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-08

CONDITIONS: Diabetic Retinopathy; Vitreous Hemorrhage Due to Diabetes Mellitus
MeSH Terms: conditions — Diabetic Retinopathy | interventions — faricimab

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Faricimab injection (Experimental): Patients will be randomized 2:1 to receive either farcimab (6 mg from 0.05 mL of a 120 mg/mL) or sham injection. The 6-mg dose of faricimab will be administered by IVT at the study site to patients. A specified filter needle must be used for each dose preparation of faricimab according to the instructions provided in the Investigator's Brochure and package insert. No other material than specified should be used. Vials of faricimab drug product are for a single-dose only (one injection preparation per patient per eye). Vials used for one patient must not be used for any other patient. Partially used vials, remaining faricimab drug product, as well as administration material must not be reused.
  Interventions: Drug: Faricimab Injection
- Sham injection (Sham Comparator): Patients will be randomized 2:1 to receive either farcimab (6 mg from 0.05 mL of a 120 mg/mL) or sham injection. The sham procedure mimics an intravitreal injection of faricimab except that the blunt end of an empty syringe is pressed against an anesthetized eye instead of a needle attached to a faricimab-filled syringe.
  Interventions: Drug: sham treatment

INTERVENTIONS:
Drug: Faricimab Injection — Pre-operative injection of bevacizumab appears to have mixed results in lowering post-operative vitreous hemorrhage. One potential reason is due to aspiration and removal of medication in the vitreous humor at the time of pars plana vitrectomy leading to less than anticipated results in controlling neovascularization and vitreous hemorrhage post-operatively. To avoid attenuation of our desired effect we plan to repeat faricimab injection post-operatively around week one.
  Other Names: Vabysmo
  Arms: Faricimab injection
Drug: sham treatment — Patients will be randomized 2:1 to receive either faricimab (6 mg from 0.05 mL of a 120 mg/mL) or sham injection
  Arms: Sham injection

SUMMARY:
In this phase IV, randomized, double-masked, sham-controlled study the investigators hope to determine the efficacy in peri-operative faricimab (Vabysmo) compared to sham in limiting complications from pars plana vitrectomy for diabetic vitreous hemorrhage with or without tractional retinal detachments.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet the following criteria for study entry:

* Signed Informed Consent Form
* Age ≥ 18 years at time of signing Informed Consent Form
* Ability to comply with the study protocol, in the investigator's judgment
* For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraception as defined below:

  * Women must remain abstinent or use contraceptive methods with a failure rate of <1% per year during the treatment period and for 3 months after the final dose of the study drug.
  * A woman is considered to be of childbearing potential if she is postmenarcheal, has not reached a postmenopausal state (≥ 12 continuous months of amenorrhea with no identified cause other than menopause), and is not permanently infertile due to surgery (i.e., removal of ovaries, fallopian tubes, and/or uterus) or another cause as determined by the investigator (e.g., Müllerian agenesis).
  * Examples of contraceptive methods with a failure rate of < 1% per year include bilateral tubal ligation, male sterilization, hormonal contraceptives that inhibit ovulation, hormone-releasing intrauterine devices, and copper intrauterine devices.
  * The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods of contraception.

Ocular inclusion criteria for study eye:

● Patients diagnosed with non-clearing vitreous hemorrhage with or without tractional retinal detachment secondary to proliferative diabetic retinopathy and undergoing pars plana vitrectomy

Exclusion Criteria:

General:

Patients who meet any of the following general exclusion criteria will be excluded from study entry:

* Any known hypersensitivity to any of the components in the faricimab injection
* Any known hypersensitivity to any dilating eye drops, disinfectants (e.g., iodine), or any of the anesthetics and antimicrobial preparations used during the study
* History of other diseases, other non-diabetic metabolic dysfunction, physical examination finding, or historical or current clinical laboratory finding giving reasonable suspicion of a condition that contraindicates the use of the faricimab or that might affect interpretation of the results of the study or renders the patient at high-risk for treatment complications, in the opinion of the investigator
* Pregnant or breastfeeding, or intending to become pregnant during the study or within 3 months after the final dose of faricimab Women of childbearing potential must have a negative urine pregnancy test result at baseline prior to initiation of dosing of faricimab/sham and a negative urine pregnancy test at post-op Week 1 prior to dosing of faricimab/sham

Ocular exclusion criteria for study eye:

Patients who meet any of the following exclusion criteria for the study eye will be excluded from study entry:

* Any ocular anti-VEGF treatment within 3 months prior to Day 1 (Baseline) in the study eye
* Vitreous hemorrhage or tractional retinal detachment suspected due to cause other than diabetic retinopathy
* Any glaucoma surgery in the study eye prior to the Day 1 (Baseline) visit
* History of vitreoretinal surgery/pars plana vitrectomy, corneal transplant, or radiotherapy in study eye
* Uncontrolled glaucoma (e.g., progressive loss of visual fields or defined as intraocular pressure (IOP) ≥25 mmHg at the Day 1 (Baseline) visit despite treatment with anti-glaucoma medication)
* Any history of idiopathic, infectious, or noninfectious uveitis
* Any current or history of ocular disease other than diabetic retinopathy that may confound assessment of the macula or affect central vision (e.g., age-related macular degeneration, retinal vein occlusion, angioid streaks, histoplasmosis, active or inactive cytomegalovirus retinitis, pathological myopia, retinal detachment, macular traction, retinal embolus, macular hole)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-07-12 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Rates of post-operative vitreous hemorrhage | 6 months
  Following treatment and surgery, the development of vitreous hemorrhage will be quantified and evaluated.

SECONDARY OUTCOMES:
BCVA outcomes | 6 and 12 months
  Vision will be tested following treatment and surgery on the Snellen Chart, with or without correction as indicated.
Rates of re-operation for non-clearing vitreous hemorrhage | 6 and 12 months
  Following treatment and surgery, if re-operation for non-clearing vitreous hemorrhage is indicated, this will be track and quantified.
Rate of post-operative epiretinal membrane formation. | Through study completion, an average of 1 year
  Following treatment and surgery, the duration of time if a patient was to develop an epiretinal membrane will be quantified and evaluated.
Rate of post-operative rhegmatogenous or tractional retinal detachment. | Through study completion, an average of 1 year
  Following treatment and surgery, the duration of time if a patient was to develop a rhegmatogenous or tractional retinal detachment will be quantified and evaluated.
Duration of operative time. | intra-operatively
  The official duration of surgical time will be quantified and evaluated.
Number of endodiathermy use exchanges intra-operatively. | intra-operatively
  At the time of surgery, the number of endodiathermy use exchanges will be counted and evaluated.
Number of retinal breaks intra-operatively. | intra-operatively
  At the time of surgery, the number of retinal breaks intra-operatively will be counted and evaluated.
Number of patients with intra-operative bleeding | intra-operatively
  At the time of surgery, the number of patients who experience intra-operative bleeding will be counted and evaluated.

CONTACTS AND LOCATIONS:
Locations (1):
- Sue Anschutz-Rodgers Eye Center, Aurora, Colorado, United States